CLINICAL TRIAL: NCT06583954
Title: PROOF OF CONCEPT OF A NEW DEVICE FOR SUBJECTIVE REFRACTION WITH LIGHTFIELD TECHNOLOGY
Brief Title: SUBJECTIVE REFRACTION WITH LIGHTFIELD TECHNOLOGY
Status: Completed | Type: Observational
Sponsor: Daniela Nosch (Other)
Responsible Party: Sponsor-Investigator, Daniela Nosch, Lecturer, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Other Study IDs: 2024-D0081; 2024-D0081 (Registry Identifier: Swissethics)
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Refractive Error Correction
Keywords: subjective refraction; phoropter; lightfield technology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- healthy adults with refractive error

SUMMARY:
The aim of this study is to test whether it is possible in principle to determine defective vision using light field technology. The measurements with this first prototype will be compared with the results of the conventional method for subjective refraction determination and those using a phoropter (Vision R-800 phoropter).

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Best corrected visual acuity ≥ 0.8 (logMAR ≤ 0.1).
* Dioptric range for hypermetropia: ≤ +4.50 D.
* Dioptric range for myopia: ≥ -6.50 D.
* Dioptric range for cylinder: ≤ -2.00 D.
* Good general health, i.e.no systemic disease such as diabetes or rheumatism which could influence ocular health
* No ocular pathology or history of (intra)ocular surgery except for cataract surgery

Exclusion Criteria:

* • Contact lens wear during the days of visit

  * Binocular vision problems (e.g. amblyopia, strabismus).
  * Inability to follow the procedures of the investigation, such as language problems, psychological disorders and dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults with refractive error
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
precision of determination of refractive error | within one week
  To explore if this prototype CREAL device based on LightField Technology can determine the refractive error reliably, in comparison to well-established methods such as subjective refraction with a trial frame and with the phoropter Vision-R 800 (Essilor SA).

SECONDARY OUTCOMES:
repeatability of all three methods for subjective refraction | within one week

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Institute of Optometry, FHNW, Olten, Canton of Solothurn
  - Insititute of Optometry, FHNW University of Applied Sciences and Arts Northwestern Switzerland, Olten

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkataraman AP, Sirak D, Brautaset R, Dominguez-Vicent A. Evaluation of the Performance of Algorithm-Based Methods for Subjective Refraction. J Clin Med. 2020 Sep 29;9(10):3144. doi: 10.3390/jcm9103144. PMID 33003297
- See also: Related Info — https://creal.com/